CLINICAL TRIAL: NCT05349045
Title: Containing Angiogenesis Inhibitor Plus Anti-PD-1/PD-L1 Antibody in Anti-tumor Treatment of Chinese Patients With Unresectable Locally Advanced / Recurrent or Metastatic Esophageal Cancer: a Real World Study
Brief Title: Angiogenesis Inhibitor Plus Anti-PD-1/PD-L1 Antibody in Advanced Esophageal Cancer
Acronym: AIPAAIAEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2022-KY-0179-002
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- an anti-PD-1/PD-L1 antibody with an angiogenesis inhibitor group
  Interventions: Drug: an anti-PD-1/PD-L1 antibody plus an angiogenesis inhibitor

INTERVENTIONS:
Drug: an anti-PD-1/PD-L1 antibody plus an angiogenesis inhibitor — This is an observational study

SUMMARY:
The combination of an anti-PD-1/PD-L1 antibody with an angiogenesis inhibitor has shown efficacy in many cancers.The purpose of this study is to confirm that the combination of these two drugs can benefit patients with advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal cancer confirmed by histopathology or cytology
2. Unresectable locally advanced/recurrent or metastatic esophageal cancer, or progression after neoadjuvant or adjuvant therapy
3. Esophageal cancer patients who benefit from the use of an anti-PD-1/PD-L1 antibody with an angiogenesis inhibitor evaluated by the researchers
4. Patients who sign informed consent and voluntarily join the study

Exclusion Criteria:

1. Patients who are recommended not using an anti-PD-1/PD-L1 antibody or an angiogenesis inhibitor in the instructions, or other patients who are judged by the investigators to be unsuitable in the study
2. Patients who are undergoing treatment regimen of blind trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Esophageal cancer confirmed by histopathology or cytology
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-05 (Estimated); Primary Completion 2024-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of admission until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | From date of admission until the date of death from any cause, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No